CLINICAL TRIAL: NCT01188772
Title: A Multi-center, Placebo-Controlled, Dose Ranging Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Following Oral Administration of PSI-7977 in Combination With Pegylated Interferon and Ribavirin in Treatment-Naïve Patients With Chronic HCV Infection Genotype 1, and an Open Label Assessment of PSI-7977 in Patients With HCV Genotypes 2 or 3
Brief Title: Sofosbuvir in Combination With Pegylated Interferon and Ribavirin and in Treatment-Naive Hepatitis C-infected Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P7977-0422
Record Dates: First submitted 2010-08-23; First posted 2010-08-25 (Estimated); Results first posted 2014-02-19 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Hepatitis C Virus
Keywords: Hepatitis C Virus; HCV; hepatitis; Genotype 1; Genotype 2; Genotype 3
MeSH Terms: conditions — Hepatitis C; Hepatitis | interventions — Sofosbuvir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Sofosbuvir 200 mg (Genotype 1) (Experimental): Participants with genotype 1 HCV infection were randomized to receive sofosbuvir 200 mg (2 x 100 mg tablets)+placebo to match sofosbuvir (2 tablets)+PEG+RBV for 12 weeks followed by PEG+RBV for up to an additional 36 weeks.
  Interventions: Drug: Sofosbuvir; Drug: Placebo to match sofosbuvir; Drug: PEG; Drug: RBV
- Sofosbuvir 400 mg (Genotype 1) (Experimental): Participants with genotype 1 HCV infection were randomized to receive sofosbuvir 400 mg (4 x 100 mg tablets)+PEG+RBV for 12 weeks followed by PEG+RBV for up to an additional 36 weeks.
  Interventions: Drug: PEG; Drug: RBV
- Placebo (Genotype 1) (Active Comparator): Participants with genotype 1 HCV infection were randomized to receive placebo to match sofosbuvir (4 tablets)+PEG+RBV for 12 weeks followed by PEG+RBV for up to an additional 36 weeks.
  Interventions: Drug: Placebo to match sofosbuvir; Drug: PEG; Drug: RBV
- Sofosbuvir 400 mg (Genotype 2/3) (Experimental): Participants with genotype 2 or 3 HCV infection received sofosbuvir 400 mg (4 x 100 mg tablets)+PEG+RBV for 12 weeks.
  Interventions: Drug: Sofosbuvir; Drug: PEG; Drug: RBV

INTERVENTIONS:
Drug: Sofosbuvir — Sofosbuvir tablets were administered orally once daily.
  Other Names: Sovaldi®; GS-7977; PSI-7977
  Arms: Sofosbuvir 200 mg (Genotype 1); Sofosbuvir 400 mg (Genotype 2/3)
Drug: Placebo to match sofosbuvir — Placebo tablets to match sofosbuvir were administered orally once daily.
  Arms: Placebo (Genotype 1); Sofosbuvir 200 mg (Genotype 1)
Drug: PEG — Pegylated interferon alfa-2a (PEG) 180 μg was administered once weekly by subcutaneous injection.
  Other Names: Pegasys®
Drug: RBV — Ribavirin (RBV) was administered as a tablet orally according to package insert dosing recommendations (Genotype 1: < 75kg = 1000 mg and ≥ 75 kg = 1200 mg; Genotype 2/3: 800 mg).
  Other Names: Copegus®

SUMMARY:
Genotype 1: Participants with genotype 1 hepatitis C (HCV) infection were randomized to receive sofosbuvir (GS-7977; PSI-7977) 200 mg or 400 mg, or matching placebo, plus pegylated interferon alfa 2a (PEG) and ribavirin (RBV) for 12 weeks, followed by PEG+RBV for an up to an additional 36 weeks. Randomization was stratified by IL28B status (CC, CT, TT) and HCV RNA level (< 800,000 IU/ml or ≥ 800,000 IU/ml) at baseline. Participants were randomized in a 2:2:1 manner; those who achieved an extended rapid virologic response (eRVR) (HCV RNA < lower limit of detection [15 IU/mL] from Weeks 4 through 12) received an additional 12 weeks of PEG+RBV. Subjects not achieving eRVR received an additional 36 weeks of PEG+RBV.

Genotype 2 and 3: Participants with genotype 2 or 3 hepatitis C (HCV) received sofosbuvir 400 mg plus PEG+RBV for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18 to 70 years, inclusive, at screening
* Documented chronic genotype 1, 2, or 3 HCV infection
* No previous treatment with HCV antiviral mediations
* Body mass index (BMI) of greater than 18 kg/m2, but not exceeding 36 kg/m2.
* Liver biopsy obtained within 3 years prior to the Day 1 visit, with a fibrosis classification of non-cirrhotic as judged by a local pathologist
* Willing to refrain from beginning any new exercise regimens during the first 3 months of the study
* Fasting blood glucose ≤ 300 mg/dl and/or glycosylated hemoglobin (HbA1c) ≤ 8
* History of hypertension only if managed effectively on a stable regimen of two or fewer antihypertensives for at least three (3) months prior to screening

Exclusion Criteria:

* Females who were breastfeeding
* Males and females of reproductive potential who are unwilling to use an "effective", protocol-specified method(s) of contraception during the study
* Positive test at Screening for HBsAg, anti-HBc IgM Ab, or anti-HIV Ab.
* History of any other clinically significant chronic liver disease
* Treatment with herbal/natural remedies with antiviral activity within 30 days prior to baseline.
* Significant history of immunologically mediated disease, cardiac or pulmonary disease, seizure disorder or anticonvulsant use
* History of ascites, variceal hemorrhage, hepatic encephalopathy, or conditions consistent with decompensated liver disease
* Use of medications associated with QT prolongation within 30 days prior to dosing
* Screening electrocardiogram (ECG) QTc value greater than 450 ms and/or clinically significant ECG findings
* Personal or family history of Torsade de pointes.
* Positive results for drugs of abuse test at screening
* Abnormal hematological and biochemical parameters, including alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 5 times the upper limit of the normal range (ULN)
* History of major organ transplantation with an existing functional graft
* History of uncontrolled thyroid disease or abnormal thyroid-stimulating hormone (TSH) levels at screening
* Clinically significant drug allergy to nucleoside/nucleotide analogs
* History or current evidence of psychiatric illness, immunologic disorder, pulmonary, cardiac disease, seizure disorder, cancer or history of malignancy that in the opinion of the investigator makes the patient unsuitable for the study
* History of systemic antineoplastic or immunomodulatory treatment within 6 months prior to dosing, or the expectation of such treatment during the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2010-08; Primary Completion 2011-04 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert H. Hyland, DPhil, Study Director — Gilead Sciences
Locations (23):
- United States (22):
  - Alabama Liver and Digestive Specialists, Montgomery, Alabama
  - Advanced Clinical Research Institute, Anaheim, California
  - SCTI Research Foundation, Coronado, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Dr. Jay Lalezari, San Francisco, California
  - Dr. Natalie Bzowej, San Francisco, California
  - Dr. David Nelson, Gainesville, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Gastrointestinal Specialists of Georgia, Marietta, Georgia
  - University of Chicago, Chicago, Illinois
  - Dr. Mark Sulkowski, Lutherville, Maryland
  - Liver Research Center Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Kansas City Gastroenterology and Hepatology, Kansas City, Missouri
  - Dr. Bruce Bacon, St Louis, Missouri
  - North Shore University Hospital, Manhasset, New York
  - Dr. Ira Jacobson, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Dr. Jama Darling, Chapel Hill, North Carolina
  - Dr. Raj Reddy, Philadelphia, Pennsylvania
  - Columbia Gastroenterology and Liver Associates, Columbia, South Carolina
  - Dr. Eric Lawitz, San Antonio, Texas
  - Digestive Disease Institute Virginia Mason Medical Center, Seattle, Washington
- Fundacion de Investigacion de Diego, Santurce, Puerto Rico, Puerto Rico

REFERENCES:
- [Derived] Lawitz E, Lalezari JP, Hassanein T, Kowdley KV, Poordad FF, Sheikh AM, Afdhal NH, Bernstein DE, Dejesus E, Freilich B, Nelson DR, Dieterich DT, Jacobson IM, Jensen D, Abrams GA, Darling JM, Rodriguez-Torres M, Reddy KR, Sulkowski MS, Bzowej NH, Hyland RH, Mo H, Lin M, Mader M, Hindes R, Albanis E, Symonds WT, Berrey MM, Muir A. Sofosbuvir in combination with peginterferon alfa-2a and ribavirin for non-cirrhotic, treatment-naive patients with genotypes 1, 2, and 3 hepatitis C infection: a randomised, double-blind, phase 2 trial. Lancet Infect Dis. 2013 May;13(5):401-8. doi: 10.1016/S1473-3099(13)70033-1. Epub 2013 Mar 15. PMID 23499158

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled in a total of 22 study sites in the United States. The first participant was screened on 16 August 2010. The last participant observation was on 11 May 2012.
Pre-assignment Details: 147 participants were randomized, and 146 participants received at least one dose of study drug, and comprise the Safety Analysis Set.
Groups:
- Sofosbuvir 200 mg (Genotype 1): Participants with genotype 1 HCV infection were randomized to receive sofosbuvir 200 mg (2 x 100 mg tablets)+placebo to match sofosbuvir (2 tablets)+pegylated interferon alfa-2a (PEG)+ribavirin (RBV) for 12 weeks followed by PEG+RBV for up to an additional 36 weeks.
Period: Overall Study
Arm/Group | Sofosbuvir 200 mg (Genotype 1) | Sofosbuvir 400 mg (Genotype 1) | Placebo (Genotype 1) | Sofosbuvir 400 mg (Genotype 2/3)
Started | 48 | 48 | 26 | 25
Randomized and Treated | 48 | 47 | 26 | 25
Completed | 43 | 45 | 15 | 24
Not Completed | 5 | 3 | 11 | 1
Not completed — Randomized but Not Treated | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 2 | 0
Not completed — Lost to Follow-up | 4 | 1 | 1 | 1
Not completed — Non-responder | 0 | 0 | 3 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Terminated by Sponsor | 0 | 0 | 1 | 0
Not completed — Treatment Failure | 0 | 0 | 1 | 0
Not completed — Virologic Failure | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who were randomized and at least one dose of study drug
Groups:
- Sofosbuvir 200 mg (Genotype 1): Sofosbuvir 200 mg+PEG+RBV for 12 weeks; PEG+RBV for up to an additional 36 weeks
- Sofosbuvir 400 mg (Genotype 1): Sofosbuvir 400 mg+PEG+RBV for 12 weeks; PEG+RBV for up to an additional 36 weeks
- Placebo (Genotype 1): Placebo to match sofosbuvir+PEG+RBV for 12 weeks; PEG+RBV for up to an additional 36 weeks
- Sofosbuvir 400 mg (Genotype 2/3): Sofosbuvir 400 mg+PEG+RBV for 12 weeks
- Total: Total of all reporting groups
Arm/Group | Sofosbuvir 200 mg (Genotype 1) | Sofosbuvir 400 mg (Genotype 1) | Placebo (Genotype 1) | Sofosbuvir 400 mg (Genotype 2/3) | Total
Number analyzed (Participants) | 48 | 47 | 26 | 25 | 146
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.4 (11.49) | 51.4 (9.37) | 48.6 (9.35) | 47.2 (11.07) | 49.2 (10.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 26 | 7 | 9 | 57
  Male | 33 | 21 | 19 | 16 | 89
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 1 | 8 | 20
  Not Hispanic or Latino | 43 | 41 | 24 | 17 | 125
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska native | 0 | 1 | 0 | 0 | 1
  Asian | 1 | 0 | 0 | 0 | 1
  Black or African American | 6 | 7 | 5 | 4 | 22
  Other | 2 | 2 | 0 | 1 | 5
  White | 39 | 37 | 21 | 20 | 117
Hepatitis C (HCV) RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.54 (0.630) | 6.39 (0.827) | 6.50 (0.762) | 6.07 (0.794) | 6.40 (0.760)
Liver Biopsy Fibrosis Score [Number; unit: participants]
  None or Minimal Fibrosis | 12 | 7 | 3 | 7 | 29
  Portal Fibrosis | 35 | 38 | 21 | 18 | 112
  Bridging Fibrosis | 1 | 2 | 2 | 0 | 5
  Cirrhosis | 0 | 0 | 0 | 0 | 0
Alanine Aminotransferase (ALT) [Mean (Standard Deviation); unit: IU/L] | 81.9 (66.07) | 76.1 (67.56) | 81.4 (49.14) | 74.5 (54.81) | 78.7 (61.53)
IL28b Genotype [Number; unit: participants] — CC, CT, and TT alleles are different forms of the IL28b gene.
  participants
    CC | 21 | 18 | 11 | 7 | 57
    CT | 24 | 19 | 11 | 17 | 71
    TT | 3 | 10 | 4 | 1 | 18

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced Adverse Events During the Sofosbuvir Treatment Period
Description: Adverse events (AEs) occurring during the sofosbuvir treatment period and for 30 days following the last dose of sofosbuvir were summarized across the participant population. A participant was counted once if they had a qualifying event.
Time Frame: Baseline to Week 12 plus 30 days
Population: Safety Analysis Set: participants were randomized and received at least one dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | Sofosbuvir 200 mg (Genotype 1) | Sofosbuvir 400 mg (Genotype 1) | Placebo (Genotype 1) | Sofosbuvir 400 mg (Genotype 2/3)
Number analyzed (Participants) | 48 | 47 | 26 | 25
percentage of participants
  Any AE | 97.9 | 97.9 | 100.0 | 96.0
  Drug-related AE | 97.9 | 95.7 | 100.0 | 96.0
  Grade 3 or higher AE | 10.4 | 21.3 | 11.5 | 12.0
  AE leading to drug discontinuation | 4.2 | 6.4 | 11.5 | 0.0
  Serious AE | 2.1 | 6.4 | 3.8 | 0.0

2. Secondary Outcome: Change in HCV RNA From Baseline to Week 12
Time Frame: Baseline to Week 12
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Sofosbuvir 200 mg (Genotype 1) | Sofosbuvir 400 mg (Genotype 1) | Placebo (Genotype 1) | Sofosbuvir 400 mg (Genotype 2/3)
Number analyzed (Participants) | 48 | 43 | 26 | 24
log10 IU/mL | -5.39 (0.630) | -5.20 (0.842) | -4.16 (1.728) | -4.95 (0.803)

3. Secondary Outcome: Percentage of Participants With Rapid Virologic Response at Week 4
Description: Rapid virologic response was defined as HCV RNA below the limit of detection (< 15 IU/mL) at Week 4 (Day 29)
Time Frame: Week 4
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Sofosbuvir 200 mg (Genotype 1) | Sofosbuvir 400 mg (Genotype 1) | Placebo (Genotype 1) | Sofosbuvir 400 mg (Genotype 2/3)
Number analyzed (Participants) | 48 | 47 | 26 | 25
percentage of participants | 97.9 | 97.9 | 19.2 | 96.0

4. Secondary Outcome: Percentage of Participants With Complete Early Virologic Response at Week 12
Description: Complete early virologic response was defined as HCV RNA below the limit of detection (< 15 IU/mL) at Week 12
Time Frame: Week 12
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Sofosbuvir 200 mg (Genotype 1) | Sofosbuvir 400 mg (Genotype 1) | Placebo (Genotype 1) | Sofosbuvir 400 mg (Genotype 2/3)
Number analyzed (Participants) | 48 | 47 | 26 | 25
percentage of participants | 100.0 | 91.5 | 61.5 | 96.0

5. Secondary Outcome: Percentage of Participants With Extended Rapid Virologic Response
Description: Extended rapid virologic response was defined as HCV RNA below the limit of detection (< 15 IU/mL) at Week 4 (Day 29) which was maintained through Week 12.
Time Frame: Week 4 to Week 12
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Sofosbuvir 200 mg (Genotype 1) | Sofosbuvir 400 mg (Genotype 1) | Placebo (Genotype 1) | Sofosbuvir 400 mg (Genotype 2/3)
Number analyzed (Participants) | 48 | 47 | 26 | 25
percentage of participants | 97.9 | 91.5 | 19.2 | 96.0

6. Secondary Outcome: Percentage of Participants With Virologic Response at the End of Treatment
Description: End-of-treatment virologic response was defined as HCV RNA below the limit of detection (< 15 IU/mL) at the last on-treatment visit.
Time Frame: Week 48 (genotype 1) or Week 12 (genotype 2/3)
Population: Participants in the Safety Analysis Set with available data were analyzed. One participant in the Sofosbuvir 400 mg (Genotype 2/3) Group was lost to follow up before the end of treatment and is not included in this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Sofosbuvir 200 mg (Genotype 1) | Sofosbuvir 400 mg (Genotype 1) | Placebo (Genotype 1) | Sofosbuvir 400 mg (Genotype 2/3)
Number analyzed (Participants) | 48 | 47 | 26 | 24
percentage of participants | 93.8 | 100.0 | 61.5 | 100.0

7. Secondary Outcome: Percentage of Participants With Sustained Virologic Response at Post-treatment Week 12 (SVR12) and 24 (SVR24)
Description: SVR12 and SVR24 were defined as HCV RNA below the limit of detection (< 15 IU/mL) at post-treatment Weeks 12 and 24, respectively.
Time Frame: Post-treatment Weeks 12 and 24
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Sofosbuvir 200 mg (Genotype 1) | Sofosbuvir 400 mg (Genotype 1) | Placebo (Genotype 1) | Sofosbuvir 400 mg (Genotype 2/3)
Number analyzed (Participants) | 48 | 47 | 26 | 25
percentage of participants
  SVR12 | 89.6 | 91.5 | 57.7 | 92.0
  SVR24 | 89.6 | 91.5 | 57.7 | 92.0

8. Secondary Outcome: Plasma Pharmacokinetics of GS-331007 (Cmax at Day 8)
Description: The pharmacokinetics of sofosbuvir metabolite GS-331007 were analyzed as the maximum observed concentration of drug in plasma (Cmax) at Day 8. Blood samples were collected at 1, 2, and 4 hours postdose for all participants, and at 8 and 12 hours postdose for participants enrolled at selected sites.
Time Frame: 1, 2, 4, 8, and 12 hours postdose
Population: Participants who had measurements of pharmacokinetic parameters at Day 8 were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Sofosbuvir 200 mg (Genotype 1): Sofosbuvir 200 mg+PEG+RBV for 12 weeks; PEG+RBV for 36 additional weeks
- Sofosbuvir 400 mg (Genotype 1): Sofosbuvir 400 mg+PEG+RBV for 12 weeks; PEG+RBV for 36 additional weeks
Arm/Group | Sofosbuvir 200 mg (Genotype 1) | Sofosbuvir 400 mg (Genotype 1) | Sofosbuvir 400 mg (Genotype 2/3)
Number analyzed (Participants) | 3 | 3 | 4
ng/mL | 331.48 (167.31) | 750.78 (108.01) | 518.18 (212.19)

9. Secondary Outcome: Plasma Pharmacokinetics of GS-331007 (Cmax at Day 15)
Description: The pharmacokinetics of sofosbuvir metabolite GS-331007 were analyzed as the Cmax at Day 15. Blood samples were collected at 1, 2, and 4 hours postdose for all participants, and at 8 and 12 hours postdose for participants enrolled at selected sites.
Time Frame: 1, 2, 4, 8, and 12 hours postdose
Population: Participants who had measurements of pharmacokinetic parameters at Day 15 were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sofosbuvir 200 mg (Genotype 1) | Sofosbuvir 400 mg (Genotype 1) | Sofosbuvir 400 mg (Genotype 2/3)
Number analyzed (Participants) | 4 | 1 | 5
ng/mL | 269.93 (65.71) | 1087.21 (NA) — Standard deviation not available as n = 1 | 515.13 (178.60)

10. Secondary Outcome: Plasma Pharmacokinetics of GS-331007 (Cmax at Day 29)
Description: The pharmacokinetics of sofosbuvir metabolite GS-331007 were analyzed as the Cmax at Day 29. Blood samples were collected at 1, 2, and 4 hours postdose for all participants, and at 8 and 12 hours postdose for participants enrolled at selected sites.
Time Frame: 1, 2, 4, 8, and 12 hours postdose
Population: Participants who had measurements of pharmacokinetic parameters at Day 29 were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sofosbuvir 200 mg (Genotype 1) | Sofosbuvir 400 mg (Genotype 1) | Sofosbuvir 400 mg (Genotype 2/3)
Number analyzed (Participants) | 5 | 2 | 5
ng/mL | 285.77 (91.43) | 897.41 (187.80) | 574.13 (241.39)

11. Secondary Outcome: Plasma Pharmacokinetics of GS-331007 (AUCtau at Day 8)
Description: The pharmacokinetics of sofosbuvir metabolite GS-331007 were analyzed as the the area under the plasma concentration versus time curve over the dosing interval (AUCtau) at Day 8. Blood samples were collected at 1, 2, and 4 hours postdose for all participants, and at 8 and 12 hours postdose for participants enrolled at selected sites.
Time Frame: 1, 2, 4, 8, and 12 hours postdose
Population: Participants who had measurements of pharmacokinetic parameters at Day 8 were analyzed.
Measure: Mean (Standard Deviation); unit: ng•h/mL
Arm/Group | Sofosbuvir 200 mg (Genotype 1) | Sofosbuvir 400 mg (Genotype 1) | Sofosbuvir 400 mg (Genotype 2/3)
Number analyzed (Participants) | 3 | 3 | 4
ng•h/mL | 3020.30 (1290.59) | 8620.07 (1717.44) | 5738.61 (2009.44)

12. Secondary Outcome: Plasma Pharmacokinetics of GS-331007 (AUCtau at Day 15)
Description: The pharmacokinetics of sofosbuvir metabolite GS-331007 were analyzed as the the area under the plasma concentration versus time curve over the dosing interval (AUCtau) at Day 15. Blood samples were collected at 1, 2, and 4 hours postdose for all participants, and at 8 and 12 hours postdose for participants enrolled at selected sites.
Time Frame: 1, 2, 4, 8, and 12 hours postdose
Population: Participants who had measurements of pharmacokinetic parameters at Day 15 were analyzed.
Measure: Mean (Standard Deviation); unit: ng•h/mL
Arm/Group | Sofosbuvir 200 mg (Genotype 1) | Sofosbuvir 400 mg (Genotype 1) | Sofosbuvir 400 mg (Genotype 2/3)
Number analyzed (Participants) | 4 | 1 | 5
ng•h/mL | 3178.53 (1179.46) | 11245.43 (NA) — Standard deviation not available as n = 1 | 5465.41 (1070.93)

13. Secondary Outcome: Plasma Pharmacokinetics of GS-331007 (AUCtau at Day 29)
Description: The pharmacokinetics of sofosbuvir metabolite GS-331007 were analyzed as the the area under the plasma concentration versus time curve over the dosing interval (AUCtau) at Day 29. Blood samples were collected at 1, 2, and 4 hours postdose for all participants, and at 8 and 12 hours postdose for participants enrolled at selected sites.
Time Frame: 1, 2, 4, 8, and 12 hours postdose
Population: Participants who had measurements of pharmacokinetic parameters at Day 29 were analyzed.
Measure: Mean (Standard Deviation); unit: ng•h/mL
Arm/Group | Sofosbuvir 200 mg (Genotype 1) | Sofosbuvir 400 mg (Genotype 1) | Sofosbuvir 400 mg (Genotype 2/3)
Number analyzed (Participants) | 5 | 2 | 5
ng•h/mL | 2789.62 (931.47) | 9191.86 (2388.88) | 5874.52 (1535.60)

14. Secondary Outcome: Percentage of Participants Who Developed Resistance to Sofosbuvir
Description: Resistance monitoring was completed in all subjects who received sofosbuvir and who had non-response, viral rebound, virologic breakthrough, or HCV RNA plateaus between Day 0 and Week 24.
Time Frame: Baseline to Week 12
Population: Participants in the Safety Analysis Set who received a regimen containing sofosbuvir were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Sofosbuvir 200 mg (Genotype 1) | Sofosbuvir 400 mg (Genotype 1) | Sofosbuvir 400 mg (Genotype 2/3)
Number analyzed (Participants) | 48 | 47 | 25
percentage of participants | 0.0 | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: Baseline to last dose or sofosbovir/placebo plus 30 days
Arm/Group | Sofosbuvir 200 mg (Genotype 1) | Sofosbuvir 400 mg (Genotype 1) | Placebo (Genotype 1) | Sofosbuvir 400 mg (Genotype 2/3)
Serious Adverse Events (participants affected / at risk) | 1/48 | 3/47 | 1/26 | 0/25
Other Adverse Events (participants affected / at risk) | 47/48 | 46/47 | 26/26 | 24/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sofosbuvir 200 mg (Genotype 1) (N=48) | Sofosbuvir 400 mg (Genotype 1) (N=47) | Placebo (Genotype 1) (N=26) | Sofosbuvir 400 mg (Genotype 2/3) (N=25)
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Retinal vein occlusion (Eye disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0
Lymphangitis (Infections and infestations) | 0 | 1 | 0 | 0
Electrocardiogram ST segment elevation (Investigations) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sofosbuvir 200 mg (Genotype 1) (N=48) | Sofosbuvir 400 mg (Genotype 1) (N=47) | Placebo (Genotype 1) (N=26) | Sofosbuvir 400 mg (Genotype 2/3) (N=25)
Anaemia (Blood and lymphatic system disorders) | 11 | 8 | 7 | 3
Neutropenia (Blood and lymphatic system disorders) | 9 | 14 | 5 | 6
Eye pain (Eye disorders) | 0 | 0 | 1 | 2
Vision blurred (Eye disorders) | 3 | 4 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 3 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 4 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 11 | 2 | 1
Dry mouth (Gastrointestinal disorders) | 2 | 4 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 2 | 0
Flatulence (Gastrointestinal disorders) | 0 | 3 | 1 | 0
Nausea (Gastrointestinal disorders) | 17 | 21 | 9 | 12
Vomiting (Gastrointestinal disorders) | 5 | 7 | 2 | 5
Asthenia (General disorders) | 1 | 1 | 1 | 4
Chest pain (General disorders) | 1 | 1 | 2 | 1
Chills (General disorders) | 18 | 19 | 10 | 9
Fatigue (General disorders) | 32 | 32 | 16 | 9
Injection site reaction (General disorders) | 7 | 4 | 2 | 0
Irritability (General disorders) | 8 | 7 | 5 | 3
Malaise (General disorders) | 5 | 3 | 1 | 1
Pain (General disorders) | 14 | 12 | 8 | 4
Pyrexia (General disorders) | 12 | 10 | 2 | 4
Nasopharyngitis (Infections and infestations) | 3 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 2 | 2 | 2 | 0
Sinusitis (Infections and infestations) | 6 | 2 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 2 | 1 | 1
Urinary tract infection (Infections and infestations) | 3 | 2 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 5 | 6 | 4 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 5 | 5 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 5 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 11 | 6 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 2
Dizziness (Nervous system disorders) | 6 | 5 | 3 | 5
Dysgeusia (Nervous system disorders) | 4 | 5 | 0 | 2
Headache (Nervous system disorders) | 17 | 20 | 15 | 11
Hyperaesthesia (Nervous system disorders) | 3 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 3
Affect lability (Psychiatric disorders) | 1 | 1 | 2 | 1
Anxiety (Psychiatric disorders) | 4 | 7 | 2 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 3 | 1
Depression (Psychiatric disorders) | 7 | 5 | 3 | 2
Insomnia (Psychiatric disorders) | 9 | 15 | 9 | 4
Mood Swings (Psychiatric disorders) | 2 | 1 | 2 | 1
Sleep disorder (Psychiatric disorders) | 5 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 6 | 3 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 4 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 1 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 5 | 2 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 1 | 2 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 7 | 3 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 1 | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 5 | 3 | 3
Pruritus generalised (Skin and subcutaneous tissue disorders) | 3 | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 14 | 15 | 4 | 3
Hot flush (Vascular disorders) | 1 | 1 | 1 | 3
Hypertension (Vascular disorders) | 1 | 3 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years